CLINICAL TRIAL: NCT05027880
Title: Examination of Web-based Single-session Growth Mindset Interventions for Reducing Adolescent Anxiety: A Four-arm Cluster Randomized Controlled Trial
Brief Title: Web-based Single-session Growth Mindset Intervention for Adolescent Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSEARS20201004001-01
Record Dates: First submitted 2021-08-20; First posted 2021-08-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Anxiety Generalized
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single-session Intervention of Growth Mindset for Anxiety (SIGMA) (Experimental): The SIGMA intervention group adapts the SSI-GP protocol in two ways: (a) by introducing the growth mindset of negative emotions rather than personality and (b) providing experiential process of negative emotion change. SIGMA consists of five components: (a) an introduction to emotions and the brain for conveying a scientific understanding of emotion and growth mindset of negative emotions; (b) stories and testimonials from high-school-aged youths who described their beliefs that people's negative emotion states (e.g., anxiety, depression, and stress) are malleable, and how these mindsets influence their coping with anxiety; (c) emotion changing experience induced by short videos; (d) common questions and misconceptions about growth mindset; and (e) self-persuasion writing exercises in which the participants write notes to younger students about the growth mindset of negative emotion.
  Interventions: Behavioral: Web-based single-session growth mindset intervention for adolescent anxiety
- Single-session Intervention on growth mindset of personality (SSI-GP) (Experimental): The SSI-GP intervention group uses the intervention protocol of Project Personality. Two bilingual native English and Chinese speakers translated it into Chinese and made adaptations to better fit the local context. The SSI-GP consist of five components: (a) an introduction to the brain about the potential of neuroplasticity and behavioural change; (b) written testimonials from older, high-school-aged youths of their belief in change of personality; (c) additional vignettes written by older youths about how growth mindset of personality helped them succeed following setbacks; (d) overview of common questions and misconceptions about growth mindset; and (e) an exercise of writing notes to younger students about the malleability of people's personal traits.
  Interventions: Behavioral: Web-based single-session growth mindset intervention for adolescent anxiety
- Active control group: Support therapy (ST) (Active Comparator): The control condition is a structurally similar web-based session of supportive therapy. The goals of supportive therapy are to encourage the client to identify and express feelings and to share their emotions-both positive and negative-with close others. The ST group does not teach or emphasize specific skills or beliefs. The active control group includes the same number of activities as do the SIGMA and SSI-GP interventions. Also, to mirror the intervention groups as closely as possible, supportive therapy includes vignettes written by similar school-aged youths, who describe times when they benefited from sharing their feelings with friends or family members.
  Interventions: Behavioral: Web-based single-session growth mindset intervention for adolescent anxiety
- SIGMA-BOOSTER (Experimental): The SIGMA-BOOSTER group receives the same intervention as the SIGMA group, the only difference is that the SIGMA-BOOSTER group receives booster messages with core intervention content every 2 weeks between the 2-week post-test and the 2-month follow-up survey, that is, a total of 5 weekly booster messages are sent to the SIGMA-BOOSTER group, which will help us determine the most effective way of implementing the intervention.
  Interventions: Behavioral: Web-based single-session growth mindset intervention for adolescent anxiety

INTERVENTIONS:
Behavioral: Web-based single-session growth mindset intervention for adolescent anxiety — This proposed study uses a four-arm, parallel group, cluster randomized controlled trial design to evaluate the efficacy of SIGMA compared to a web-based growth mindset SSI (SSI-GP) and an active web-based control programme. The concurrent parallel group structure assures that the different groups take part in their respective intervention at the same time.

SUMMARY:
Anxiety disorders are the most common mental disorders worldwide. In Hong Kong, 7% of adolescents are diagnosed with anxiety disorders, and one in every four secondary school students reports clinical-level anxiety symptoms. However, 65% of them do not access services. Long waitlists in public services, the high cost of private services, or the fear of being stigmatized can hinder service access. The high prevalence of anxiety and low intervention uptake indicate a pressing need to develop timely, scalable, and potent interventions suitable for adolescents. Single-session interventions (SSIs) have the potential to be scalable interventions for diagnosable or subclinical psychopathology in adolescents. Providing precise and context-adapted intervention is the key to achieving intervention efficacy. This study aims to compare the effectiveness of four SSIs: Single-session Intervention of Growth Mindset for Anxiety (SIGMA), SIGMA with booster messages, SSI of Growth mindset of Personality (SSI-GP), and active control using support therapy (ST), in reducing adolescent anxiety. Adolescents (N=731, aged 12-20) from secondary schools have been randomized to one of the four intervention conditions: the SIGMA, SIGMA-BOOSTER, SSI-GP, or active control. The implementation of each intervention is approximately 45 minutes in length. Adolescent participants reported anxiety symptoms, depression symptoms, and suicidal/self-hurting thoughts (primary outcomes); perceived control, hopelessness, attitude toward help-seeking and psychological well-being (secondary outcomes) at pre-intervention, the 2-week and 8-week follow-up. A pilot test has confirmed the feasibility and acceptability of SIGMA among adolescents. We hypothesized that SIGMA (including SIGMA and SIGMA-BOOSTER) and SSI-GP will result in a larger reduction in anxiety symptoms than the control intervention. We also predict SIGMA (including SIGMA and SIGMA-BOOSTER) will be more effective than SSI-GP. We will use the intention-to-treat principle and generalised estimating equation models for data analysis. This study was conducted from December 2022 to June 2023, with results expected to be available by March 2024. This protocol introduces the implementation content and strategies of growth mindset SSIs among school students. The study will provide evidence on the efficacy of different growth mindset SSIs for adolescent anxiety. It will also establish implementation strategies for self-administrative SSIs among school students, which can serve as a pioneer implementation of a scalable and self-accessible brief intervention to improve the well-being of young people.

ELIGIBILITY:
Inclusion Criteria:

1. secondary school students in grades 7-11;
2. Chinese youth who can read and write Chinese;
3. enough visual and auditory abilities to complete the intervention and assessment;
4. ability to give assent to participate in the study.

Exclusion Criteria:

1. no parental consent;
2. inability to stay focused to complete the intervention which is approximately 45 minutes;
3. intellectual disability or severe illness or pain that would lead to significant bias in students' health and mental health situation.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 731 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Anxiety Symptoms | baseline
  Anxiety symptoms measured by the Generalised Anxiety Disorder-7 (GAD-7) are the primary outcome. The GAD-7 scale includes seven items that assess whether anxiety symptoms have bothered the individual in the previous two weeks, ranging the frequency from 0 (not at all) to 3 (nearly every day). Example items were "Feeling nervous, anxious, or on edge", and "Not being able to stop or control worrying". GAD-7 is the self-rating scale and effectively reflects symptom severity in adolescents; it is highly correlated with clinician-administered ratings of anxiety symptoms. It is brief and suitable for self-report study. Cronbach's alpha was .93.
Anxiety Symptoms | 2-week post-intervention
  Anxiety symptoms measured by the Generalised Anxiety Disorder-7 (GAD-7) are the primary outcome. The GAD-7 scale includes seven items that assess whether anxiety symptoms have bothered the individual in the previous two weeks, ranging the frequency from 0 (not at all) to 3 (nearly every day). Example items were "Feeling nervous, anxious, or on edge", and "Not being able to stop or control worrying". GAD-7 is the self-rating scale and effectively reflects symptom severity in adolescents; it is highly correlated with clinician-administered ratings of anxiety symptoms. It is brief and suitable for self-report study. Cronbach's alpha was .93.
Anxiety Symptoms | 8-week post-intervention
  Anxiety symptoms measured by the Generalised Anxiety Disorder-7 (GAD-7) are the primary outcome. The GAD-7 scale includes seven items that assess whether anxiety symptoms have bothered the individual in the previous two weeks, ranging the frequency from 0 (not at all) to 3 (nearly every day). Example items were "Feeling nervous, anxious, or on edge", and "Not being able to stop or control worrying". GAD-7 is the self-rating scale and effectively reflects symptom severity in adolescents; it is highly correlated with clinician-administered ratings of anxiety symptoms. It is brief and suitable for self-report study. Cronbach's alpha was .93.
Depression, and suicidal/self-hurting thoughts | baseline
  The Patient Health Questionnaire-9 (PHQ-9) is used to measure participants' depression level and suicidal/self-hurting thoughts. The PHQ-9 scale includes nine items that assessed whether the depression symptoms and suicidal/self-hurting thoughts have bothered the individual in the previous two weeks, ranging the frequency from 0 (not at all) to 3 (nearly every day). Depression level is indexed by the sum of the first 8 items, while the last item indicates the suicidal/self-hurting thoughts. Example items of the PHQ-9 were "Little interest or pleasure in doing things", "Feeling down, depressed or hopeless", and "Thoughts that you would be better off dead or of hurting yourself in some way".
Depression, and suicidal/self-hurting thoughts | 2-week post-intervention
  The Patient Health Questionnaire-9 (PHQ-9) is used to measure participants' depression level and suicidal/self-hurting thoughts. The PHQ-9 scale includes nine items that assessed whether the depression symptoms and suicidal/self-hurting thoughts have bothered the individual in the previous two weeks, ranging the frequency from 0 (not at all) to 3 (nearly every day). Depression level is indexed by the sum of the first 8 items, while the last item indicates the suicidal/self-hurting thoughts. Example items of the PHQ-9 were "Little interest or pleasure in doing things", "Feeling down, depressed or hopeless", and "Thoughts that you would be better off dead or of hurting yourself in some way".
Depression, and suicidal/self-hurting thoughts | 8-week post-intervention
  The Patient Health Questionnaire-9 (PHQ-9) is used to measure participants' depression level and suicidal/self-hurting thoughts. The PHQ-9 scale includes nine items that assessed whether the depression symptoms and suicidal/self-hurting thoughts have bothered the individual in the previous two weeks, ranging the frequency from 0 (not at all) to 3 (nearly every day). Depression level is indexed by the sum of the first 8 items, while the last item indicates the suicidal/self-hurting thoughts. Example items of the PHQ-9 were "Little interest or pleasure in doing things", "Feeling down, depressed or hopeless", and "Thoughts that you would be better off dead or of hurting yourself in some way".

SECONDARY OUTCOMES:
Perceived control | baseline
  The Anxiety Control Questionnaire-Emotion Control (ACQ-EC) is a 15-item questionnaire that measures how much perceived control participants have over their anxiety. It is one of the 3 validated subscales of the Anxiety Control questionnaire, and contains 5 items (e.g., I am able to control my level of anxiety), including one reversed item (i.e., When I am anxious, I find it hard to focus on anything other than my anxiety), rated from 0 (strongly disagree) to 5 (strongly agree). The scale has a well-validated factor structure in a non-clinically selected sample, is strongly associated with anxiety and depression symptoms, and has demonstrated good internal consistency in previous investigations. Cronbach's alpha was .73.
Perceived control | 2-week post-intervention
  The Anxiety Control Questionnaire-Emotion Control (ACQ-EC) is a 15-item questionnaire that measures how much perceived control participants have over their anxiety. It is one of the 3 validated subscales of the Anxiety Control questionnaire, and contains 5 items (e.g., I am able to control my level of anxiety), including one reversed item (i.e., When I am anxious, I find it hard to focus on anything other than my anxiety), rated from 0 (strongly disagree) to 5 (strongly agree). The scale has a well-validated factor structure in a non-clinically selected sample, is strongly associated with anxiety and depression symptoms, and has demonstrated good internal consistency in previous investigations. Cronbach's alpha was .73.
Perceived control | 8-week post-intervention
  The Anxiety Control Questionnaire-Emotion Control (ACQ-EC) is a 15-item questionnaire that measures how much perceived control participants have over their anxiety. It is one of the 3 validated subscales of the Anxiety Control questionnaire, and contains 5 items (e.g., I am able to control my level of anxiety), including one reversed item (i.e., When I am anxious, I find it hard to focus on anything other than my anxiety), rated from 0 (strongly disagree) to 5 (strongly agree). The scale has a well-validated factor structure in a non-clinically selected sample, is strongly associated with anxiety and depression symptoms, and has demonstrated good internal consistency in previous investigations. Cronbach's alpha was .73.
Hopelessness | baseline
  The four-item helplessness subscale of the Demoralization Scale will be used to measure the participants' faith in the future. Each item scores on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), and the mean of all 4 items is taken to measure the hopelessness, with a higher score meaning correspondingly higher level of hopelessness. An example item is "I feel hopeless". The Cronbach's alpha of the Chinese version of this helplessness subscale was .72.
Hopelessness | 2-week post-intervention
  The four-item helplessness subscale of the Demoralization Scale will be used to measure the participants' faith in the future. Each item scores on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), and the mean of all 4 items is taken to measure the hopelessness, with a higher score meaning correspondingly higher level of hopelessness. An example item is "I feel hopeless". The Cronbach's alpha of the Chinese version of this helplessness subscale was .72.
Hopelessness | 8-week post-intervention
  The four-item helplessness subscale of the Demoralization Scale will be used to measure the participants' faith in the future. Each item scores on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), and the mean of all 4 items is taken to measure the hopelessness, with a higher score meaning correspondingly higher level of hopelessness. An example item is "I feel hopeless". The Cronbach's alpha of the Chinese version of this helplessness subscale was .72.
Attitude towards seeking help | baseline
  We use two items from the Attitude toward Seeking Counselling Help Assessment (ATSCHA) to measure participants' understanding of counselling and attitudes toward seeking counselling help. An example item is "If I believed I was having a mental breakdown, my first inclination would be to get professional attention". Cronbach's alpha was .72. We develop a brief scale including three items to assess participants' help-seeking behaviour. The three items are "when I encounter difficulties, I will not ask help from teachers", "when I encounter difficulties, I will not ask help from social workers/counsellors", and "Professional counseling and treatments can help people improve mental health". This scale will be rated on a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
Attitude towards seeking help | 2-week post-intervention
  We use two items from the Attitude toward Seeking Counselling Help Assessment (ATSCHA) to measure participants' understanding of counselling and attitudes toward seeking counselling help. An example item is "If I believed I was having a mental breakdown, my first inclination would be to get professional attention". Cronbach's alpha was .72. We develop a brief scale including three items to assess participants' help-seeking behaviour. The three items are "when I encounter difficulties, I will not ask help from teachers", "when I encounter difficulties, I will not ask help from social workers/counsellors", and "Professional counseling and treatments can help people improve mental health". This scale will be rated on a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
Attitude towards seeking help | 8-week post-intervention
  We use two items from the Attitude toward Seeking Counselling Help Assessment (ATSCHA) to measure participants' understanding of counselling and attitudes toward seeking counselling help. An example item is "If I believed I was having a mental breakdown, my first inclination would be to get professional attention". Cronbach's alpha was .72. We develop a brief scale including three items to assess participants' help-seeking behaviour. The three items are "when I encounter difficulties, I will not ask help from teachers", "when I encounter difficulties, I will not ask help from social workers/counsellors", and "Professional counseling and treatments can help people improve mental health". This scale will be rated on a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree).
Psychological wellbeing | baseline
  The short version Warwick-Edinburgh Mental Well-being Scale (WEMWBS-14) will be used to measure the extent to which participants generally experience well-being states. The WEMWBS includes 14 items, scoring on a 5-pont Likert scale ranging from 1 (none of the time) to 5 (all of the time), the average of all 14 items indicates the well-being of the participants. Sample item is "I have been feeling optimistic about the future". Cronbach's alpha was .93.
Psychological wellbeing | 2-week post-intervention
  The short version Warwick-Edinburgh Mental Well-being Scale (WEMWBS-14) will be used to measure the extent to which participants generally experience well-being states. The WEMWBS includes 14 items, scoring on a 5-pont Likert scale ranging from 1 (none of the time) to 5 (all of the time), the average of all 14 items indicates the well-being of the participants. Sample item is "I have been feeling optimistic about the future". Cronbach's alpha was .93.
Psychological wellbeing | 8-week post-intervention
  The short version Warwick-Edinburgh Mental Well-being Scale (WEMWBS-14) will be used to measure the extent to which participants generally experience well-being states. The WEMWBS includes 14 items, scoring on a 5-pont Likert scale ranging from 1 (none of the time) to 5 (all of the time), the average of all 14 items indicates the well-being of the participants. Sample item is "I have been feeling optimistic about the future". Cronbach's alpha was .93.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu S, Hu Y, Qi D, Tse S, Chan KL, Sun J, Lee P. Effects of Web-Based Single-Session Growth Mindset Interventions for Reducing Adolescent Anxiety: Four-Armed Randomized Controlled Trial. JMIR Pediatr Parent. 2025 Apr 18;8:e63500. doi: 10.2196/63500. PMID 40249649
- [Derived] Zhu S, Tse S, Chan KL, Lee P, Cheng Q, Sun J. Examination of Web-Based Single-Session Growth Mindset Interventions for Reducing Adolescent Anxiety: Study Protocol of a 3-Arm Cluster Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 17;12:e41758. doi: 10.2196/41758. PMID 36930199